CLINICAL TRIAL: NCT03732508
Title: SHR-1316, a Novel Anti-PD-L1 Antibody, in Combination With Irinotecan Liposome and Fluorouracil in Patients With Esophageal Squamous Cell Cancer: a Phase II Study
Brief Title: SHR-1316 in Combination With Chemotherapy in Patients With Esophageal Squamous Cell Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRI-SHR-1316-201
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Advanced Esophageal Squamous Cell Cancer
MeSH Terms: interventions — irinotecan sucrosofate; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan liposome plus SHR1316 plus fluorouracil (Experimental)
  Interventions: Drug: Irinotecan liposome; Drug: SHR-1316; Drug: Fluorouracil

INTERVENTIONS:
Drug: Irinotecan liposome — Irinotecan liposome intravenous infusion will be administered during the first day of treatment.
Drug: SHR-1316 — SHR-1316 intravenous infusion will be administered during the first day of treatment.
Drug: Fluorouracil — Fluorouracil intravenous infusion will be administered during the first day of treatment.

SUMMARY:
The purpose of this study is to evaluate the progression-free survival (PFS) of Chemotherapy combined with SHR-1316 in patients with advanced esophageal squamous cell cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed unresectable local advanced/recurrent or metastasis esophageal squamous cell carcinoma;
2. No previous systemic anti-tumor treatment;
3. Subjects must have at least one measurable tumor lesion per RECIST 1.1;
4. ECOG: 0-1;
5. Adequate organ and bone marrow function;

Exclusion Criteria:

1. Allergic to monoclonal antibodies, any SHR-1316 components,Irinotecan , Fluorouracil ;
2. Prior therapy as follow:

   1. Anti-PD-1 or anti-PD-L1;
   2. Any experimental drugs within 4 weeks of the first dose of study medication;
   3. Received major operations or serious injuries within 4 weeks of the first dose of study medication;
   4. Received last dose of anticancer therapy (including chemotherapy, radiotherapy, targeted therapy, etc.) within 4 weeks of the first dose of study medication;
3. Not recovered to ≤CTCAE 1 from adverse events (except for hair loss) due to a previously anti-tumor treatment;
4. Subjects with any active autoimmune disease or history of autoimmune disease;
5. Pregnancy or breast feeding;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Duration of Progression-Free Survival (PFS) | approximately 22 months
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | approximately 22 months
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
Objective Response Rate(ORR) | approximately 22 months
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
Overall Survival(OS) | approximately 22 months
  OS is defined as the time from registration to death due to any cause, or censored at date last known alive.
Adverse Events(AE) | approximately 22 months
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital,Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No